CLINICAL TRIAL: NCT03419546
Title: Clinical Validation Trial of the Single-use Bronchoscope Ambu® aScope ™ 4
Brief Title: Clinical Validation Trial of a Single-use Bronchoscope (Ambu® aScope ™ 4)
Status: Completed | Type: Observational
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Ambu A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: EO 131/2017_FJD
Record Dates: First submitted 2018-01-19; First posted 2018-02-05 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Bronchoscopic lavage with cell analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bronchoscopic procedures: Bronchoscopies performed in different sites to evaluate the level of satisfaction of the operators with the device Ambu® aScope™ 4

SUMMARY:
The aim of this study is to evaluate the usefulness of the new Ambu® aScope ™ 4 bronchoscope, in the usual practice of low complexity diagnostic bronchoscopy managed by bronchoscopists who meet the minimum training requirements (having performed 100 supervised procedures [ 10]) and maintenance of competition (with more than 25 bronchoscopies per year [10]).

DETAILED DESCRIPTION:
Muticentric trial to evaluate three outcomes

1. Describe the experience of bronchoscopists performing low complexity bronchoscopic procedures with the Ambu® aScope ™ 4.
2. Collect the opinion of bronchoscopists about the technical characteristics of the device subject to study through a standardized questionnaire.
3. Analyze the quality of both microbiological and cytological samples obtained through the disposable bronchoscope.

ELIGIBILITY:
Inclusion Criteria:

* Low complexity bronchoscopies in patients that need to undergo a low complexity bronchoscopy in the sites of the study

Exclusion Criteria:

* No acceptance of the informed consent
* Any procedure out of a low complexity bronchoscopy in the sites of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Patients that require a low complexity bronchoscopy that accept the informed consent
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Bronchoscope Quality questionnaire evaluation | Feb 2018- july 2018
  - A numeric scale describes the experience of bronchoscopists performing low complexity bronchoscopic procedures with the Ambu® aScope ™ 4.

SECONDARY OUTCOMES:
-Opinion of the operator -Quality of the sample | Feb 2018 -july 2018
  1.A numeric scale collects the opinion of bronchoscopists about the technical characteristics of the device subject to study through a standardized questionnaire.
- Sample quality | Feb 2018- july 2018
  2.Analyze the quality of both microbiological and cytological samples obtained through the disposable bronchoscope describing the diagnostic yield.

CONTACTS AND LOCATIONS:
Overall Officials: Javier Flandes, Principal Investigator — Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Locations (1):
- Fundacion Jimenez Diaz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No